CLINICAL TRIAL: NCT05898256
Title: A Single-arm, Multicenter, Phase II Study Evaluating the Efficacy and Safety of Cadonilimab Plus Chemotherapy for Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Cadonilimab in the Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Kai Hu, professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMUHK4
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bispecific Antibody + GP Group (Experimental): Cadonilimab will be administered once every 3 weeks (Q3W), for up to 2 years；
  Gemcitabine on Day 1, Day 8 of each 3 weeks cycle, for 4 to 6 cycles；
  Cisplatin on Day 1 of each 3 weeks cycle, for 4 to 6 cycles.
  Interventions: Drug: Cadonilimab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Cadonilimab — 10mg/kg administered intravenously (IV)
  Other Names: AK104
Drug: Gemcitabine — 1 g/m2, administered as an IV infusion within 30 minutes
Drug: Cisplatin — 80 mg/m2, administered as an IV infusion over 4 hours

SUMMARY:
This study is a single-arm, multicenter clinical study to evaluate the efficacy and safety of Cadonilimab in combination with gemcitabine/cisplatin as a first-line treatment for recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form (ICF) voluntarily；
2. Age ≥18 years and ≤65 years；
3. Subjects with histopathological diagnosis of nasopharyngeal carcinoma；
4. Primarily metastatic (stage IVB as defined by AJCC staging system for NPC, eighth edition) or recurrent/metastatic NPC that is not amenable to local regional treatment or curative treatment and at least 6 months after radical treatment；
5. Has not received prior systemic treatment;
6. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
7. Subject must have a measurable target lesion based on RECIST v1.1;

Exclusion Criteria:

1. Allergic to monoclonal antibodies, any cadonilimab components, gemcitabine, cisplatin, and other platinum drugs;
2. Prior therapy as follow:

   Anti-PD-1, anti-PD-L1 or anti-CTLA-4; Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment（Except：inhalation or topical corticosteroids）.
3. Any active malignancy ≤ 2 years before randomization except for specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)；
4. Female patients who are at pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to approximately 2 years
  ORR is proportion of patients with complete response(CR) or partial response(PR) assessed by investigators according to RECIST v1.1.
Incidence and severity of adverse events(AEs) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of Cadonilimab in combination with chemotherapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the first dose of Cadonilimab until documentation of PD (as per RECIST v1.1) or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 2 years
  Overall survival (OS) is defined as the time from the first dose of Cadonilimab until death due to any cause.
Disease control rate (DCR) | Up to approximately 2 years
  DCR is proportion of patients with complete response, partial response or stable disease assessed by investigators according to RECIST v1.1.

IPD SHARING:
Plan to Share IPD: No